CLINICAL TRIAL: NCT00515333
Title: An Exploratory Placebo-Controlled, Dose-Ranging Study of the Effects of TRx0014 30 MG TID, 60 MG TID AND 100 MG TID in Patients With Mild or Moderate Dementia of the Alzheimer Type
Brief Title: TRx0014 in Patients With Mild or Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Professor Claude M. Wischik, TauRx Therapeutics Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRx-014-001
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Dementia, Alzheimer Type
Keywords: Alzheimer; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo: 0 milligrams; t.i.d.
  Interventions: Drug: Placebo
- 2 (Active Comparator): Treatment group: 30 milligrams; t.i.d.
  Interventions: Drug: TRx0014
- 3 (Active Comparator): Treatment group: 60 milligrams; t.i.d.
  Interventions: Drug: TRx0014
- 4 (Active Comparator): Treatment group: 100 milligrams; t.i.d.
  Interventions: Drug: TRx0014

INTERVENTIONS:
Drug: TRx0014 — Hard capsule; 60 milligrams; t.i.d.
  Arms: 3
Drug: TRx0014 — Hard capsule; 30 milligrams; t.i.d.
  Arms: 2
Drug: Placebo — Hard capsule; 0 milligrams; t.i.d.
  Arms: 1
Drug: TRx0014 — Hard capsule, 100 milligrams, t.i.d.
  Arms: 4

SUMMARY:
The primary objective of the study is to investigate the effects of oral TRx0014 at three doses (30, 60 and 100 mg tid) compared with placebo on cognitive ability in patients with mild or moderate dementia of the Alzheimer type. Cognitive ability will be measured by the Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog). The primary evaluation will be made at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient may be of either sex and must be supervised by a carer who is competent to ensure compliance with the medication and who is willing to participate in completing the various assessments.
* Patients must be able to give written informed consent to participate in this study. Patients who lack capacity to consent may not be entered.
* Competent carer must be available and must provide written consent to his or her own participation in the study.
* Clinical diagnosis of dementia of the Alzheimer type determined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria and a diagnosis of Probable Alzheimer's Disease determined by the National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria. Information to support the diagnosis will include that derived from:

  * an abbreviated Cambridge Mental Disorders of the Elderly Examination (short CAMDEX) schedule, performed within six weeks prior to the baseline visit (Visit 0).
  * Computerised tomography (CT) or magnetic resonance imaging (MRI), with no time limit on previous scans. In centres conducting SPECT/PET scans as part of their routine practice or as part of the study these may be used to inform the NINCDS-ADRDA diagnosis.
* Patient must have mild or moderate dementia as determined by:

  * Mini-Mental State Examination (MMSE) value at screening of between 10 and 26 inclusive.
  * Clinical Dementia Rating (CDR) at screening of Stage 1 or Stage 2.

Exclusion Criteria:

* Patient has a known sensitivity to TRx0014, similar agents or any of the excipients used.
* Screening blood sample shows that the patient has glucose-6-phosphate dehydrogenase deficiency.
* Patient has known hereditary methaemoglobinaemia, has been known to have suffered an attack of acquired methaemoglobinaemia or has a blood level of methaemoglobin at screening which is above the upper limit of normal for age and laboratory.
* Patient has significant impairment of renal, hepatic or haematological function for the age of the patient.
* Patient is currently taking other anti-dementia drugs (e.g. memantine, cholinesterase inhibitors) or has taken these within the previous six weeks.
* It is anticipated that there will be a definite indication for the commencement of other licensed anti-dementia drug treatment within the 24 week treatment period of the trial.
* Patient has started taking other medication known to have an effect on mood or cognition (e.g. anticholinergics, hypnotics, sedatives, anxiolytics, neuroleptics, antidepressants, antiepileptics) within the previous six weeks; or has changed their dose of these medications within the previous six weeks.
* Patient has started taking 'alternative therapy' for AD e.g. vitamin E, folic acid, hormone replacement therapy (HRT), ginkgo biloba within the previous six weeks; or has changed their dose of these treatments within the previous six weeks.
* Patient is receiving warfarin or digitalis or any other medication that has a narrow margin between effective dose and toxic dose or between effective dose and ineffective dose, where the subject would be at risk if the levels were elevated or fell due to interaction with TRx0014.
* Patients who are unlikely to comply with trial visit schedule or with trial medication.
* Significant intercurrent illness which may compromise safety of the patient/validity of the data.
* Females with the potential of childbearing and are not using adequate contraception or females who are breastfeeding.
* Patients with a history of alcohol and/or drug abuse, defined as meeting DSM-IV criteria for substance dependence. This applies to alcohol and/or any illicit drug, including cannabis within the last six months.
* Patient has participated in a clinical investigation of a medication or device within the previous three months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cognitive ability (ADAS-cog) | At 24 weeks

SECONDARY OUTCOMES:
Behavioural and psychological symptoms (NPI) | At 12 and 24 weeks
Global performance (ADCS-CGIC) | At 12 and 24 weeks
Dementia severity (CDR-sb) | At 12 and 24 weeks
Cognition (MMSE) | At 12 and 24 weeks
Dementia caseness (Short CAMDEX) | At 12 and 24 weeks
Cognitive function (ADAS-cog) | At 6, 12, 18 and 24 weeks
Daily activities of living (BADLS) | At 12 and 24 weeks
Changes in cerebral perfusion pattern (SPECT or PET) | At baseline and between 24-26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claude M Wischik, MBChB, Study Chair — TauRx Therapeutics Ltd; Peter Bentham, MBChB, Principal Investigator — Queen Elizabeth Psychiatric Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Wischik CM, Staff RT, Wischik DJ, Bentham P, Murray AD, Storey JM, Kook KA, Harrington CR. Tau aggregation inhibitor therapy: an exploratory phase 2 study in mild or moderate Alzheimer's disease. J Alzheimers Dis. 2015;44(2):705-20. doi: 10.3233/JAD-142874. PMID 25550228